CLINICAL TRIAL: NCT06945055
Title: Integration of a Culturally Responsive Family Peer Delivered Engagement Strategy in Coordinated Specialty Care
Brief Title: FAmily Engagement Strategy for Coordinated Specialty Care
Acronym: FAMES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Oladunni Oluwoye, Associate Professor, Washington State University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 144707-002; R01MH136132 (NIH)
Record Dates: First submitted 2025-03-24; First posted 2025-04-25 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Family Members; Implementation
Keywords: early psychosis; family peer; engagement
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: A cluster randomized stepped wedge design with an attention control condition (n=225 dyads) lasting 18 months and an active implementation condition (n=225 dyads) lasting 30 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention Control Condition (Active Comparator): 225 dyads (family members/support persons and individuals receiving services for psychosis) will be recruited over a period of 18 months to receive 12 weeks of weekly communication via text, email or phone call, which includes positive messaging, community resources, appointment reminders, and psychoeducation.
  Interventions: Behavioral: Control
- Active Condition (Active Comparator): This arm lasts for 30 months during each wave of the clustered randomized stepped wedge design. 225 participants will receive the FAMES intervention.
  Interventions: Behavioral: FAMES

INTERVENTIONS:
Behavioral: FAMES — 225 dyads (family member/support persons and individuals receiving services for psychosis) will be recruited over a period of 30 months. Family member/support persons will be connected to a family peer for a period of 12 weeks who will use the cultural formulated interview to develop rapport and identify unique cultural needs which can inform treatment and resource identification. Participants will receive brief contact, family psychoeducation, and be connected to an online family resource group where they can receive additional support from certified peers and other family member/support persons.
  Arms: Active Condition
Behavioral: Control — participants will receive 12 weeks of automated communication which contain positive messaging, appointment reminders, links to community resources, and coping skills.
  Arms: Attention Control Condition

SUMMARY:
Family members/support persons' engagement in mental health services has been linked to reduced burden and stress and improves engagement and outcomes in individuals in the early stages of psychosis. The goal of FAMES is to address low family member/support person engagement in services. FAMES will also address disparities in coordinated specialty care (CSC) by using a culturally responsive family engagement strategy to be delivered by family peers.

DETAILED DESCRIPTION:
The overall goal of this mixed-methods, clustered stepped-wedged designed study is to examine the effectiveness of a family peer implemented in coordinated specialty care programs at engaging family members in services. The use of a family peer is anticipated to increase family member participant's feelings of connectedness, self-efficacy, and motivation which will in turn improve family member participants engagement in scheduled coordinated specialty care services such as family psychoeducation.

Recruitment will consist of dyads compromised of a family member support person and a corresponding individual receiving coordinated specialty care services. Recruitment will occur over two waves, the attention control condition (ACC) and the FAMES condition. The ACC will last for 18 months and will recruit 225 participant dyads during which time family member participants will be contacted weekly for 12 weeks where they will be provided with positively framed messaging, educational materials around psychosis, tips for addressing relevant concerns in areas such as communication and de-escalation, and a list of community-based and online resources and events. The FAMES condition will last for 30 months and will recruit 225 participant dyads during which time family member participants will receive a modified cultural formulation interview, brief check-ins, psychoeducation, and will have access to an online community.

Recruitment will take place at nine coordinated specialty care programs across four states (Washington, Oregon, Tennessee, and New Mexico) which have been randomized to a clustered stepped wedge program design.

ELIGIBILITY:
Family Member / Support Person Inclusion Criteria:

* Family member/support person of an individual enrolled in coordinated specialty care services for less than or equal to 6 months.
* 18 years of age or older.
* During the active implementation period (FAMES) did not participate in the attention control condition.

Exclusion Criteria:

* If they do not understand the consent process.
* If they do not speak and/or understand English or Spanish.

Primary Service User Inclusion Criteria

* enrolled in coordinated specialty care services for less than or equal to 6 months.
* 15 years of age or older.
* Has a family member/support person willing to engage in the study. during the active implementation period (FAMES) did not participate in the attention control condition.

Exclusion Criteria

* if they do not understand the consent process
* If they do not speak and/or understand English or Spanish

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Engagement in coordinated specialty care psychoeducation | Baseline through study completion; repeated measure to assess change through study completion, average of 3 months
  Will be measured as first session attendance rate and total attendance rate per family provided by administrative data from the coordinated specialty care site partners.
Engagement in Family Engagement Strategy | Baseline through study completion; repeated measure to assess change through study completion, average of 3 months
  Total number of Family Engagement Strategy session attended and the total number of contact minutes to measure engagement.

SECONDARY OUTCOMES:
Perceived Stress Scale | Baseline through study completion; repeated measure to assess change through study completion, average of 6 months
  A self-report measure which includes 10 Likert-style items to assess the degree to which an individual appraises life as stressful. Scores range from 0-40 where scores greater that 13 indicate moderate to high perceived stress.
General Anxiety Disorder - 7 | Baseline through study completion; repeated measure to assess change through study completion, average of 6 months
  Self-report measure to assess symptoms of anxiety. Scores range from 0-21 where scores greater than 10 are indicative of clinically significant anxiety.
Client Engagement | Baseline through study completion; repeated measure to assess change through study completion, average of 6 months
  Provider reported service utilization. Total number of appointments attended.
Client - Patient Health Questionnaire - 9 | Baseline through study completion; repeated measure to assess change through study completion, average of 6 months
  A self-report from the individual receiving coordinated specialty care services on their symptoms of depression. Scores range from 0-27 where any score 10 or greater is indicative of clinically significant symptoms of depression.
Family - Patient Health Questionnaire - 9 | Baseline through study completion; repeated measure to assess change through study completion, average of 6 months
  A self-report from the family member participant on their symptoms of depression. Scores range from 0-27 where any score 10 or greater is indicative of clinically significant symptoms of depression.
Community Assessment of Psychic Experiences - Positive Scale 15-items Scale | Baseline through study completion; repeated measure to assess change through study completion, average of 6 months
  A self-report measure from the individual receiving the coordinated specialty care services. Scores range from 0-3 where scores greater than 1.46 indicate clinically significant symptoms of psychosis.

OTHER OUTCOMES:
General Self-Efficacy Scale | Baseline and Month 3 of treatment period; repeated measure to assess change through study completion, an average of 3 months
  A self-report 10-item measure completed by the family member participant. Scores range from 10-40 with higher scores indicating greater self-efficacy.
Social Connectedness subscale of the Youth Services Survey - Families | Baseline and Month 3 of treatment period; repeated measure to assess change through study completion, an average of 3 months
  Social connectedness will be measured using four questions (e.g., "I know people who will listen and understand me when I need to talk") from the YSS-F. Scores range from 4 to 20, higher scores indicating greater social connectedness.
Treatment Motivation Questionnaire | Baseline and Month 3 of treatment period; repeated measure to assess change through study completion, an average of 3 months
  A self-report measure completed by the family member/support person participant. Includes 26 Likert-scale questions to assess motivation about services. Scores range from 27 to 182 where greater scores indicated greater motivation.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Deschutes County Behavioral Health EASA, Bend, Oregon
  - Comprehensive Healthcare, Pasco, Washington
  - Lucid Living, Tacoma, Washington
  - Comprehensive Healthcare, Yakima, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oluwoye O, Stokes B, Crisanti AS, Garcia KS, Kriegel L, Puzia M, Sanchez AL, Shelton RC, Weeks DL. FAMily Motivational Engagement Strategy (FAMES) for coordinated specialty care programs: study protocol to evaluate a culturally responsive engagement intervention and equity focused implementation strategies in a hybrid type 2 randomized stepped-wedge trial. Trials. 2025 Dec 16;26(1):568. doi: 10.1186/s13063-025-09280-0. PMID 41402877